CLINICAL TRIAL: NCT00219726
Title: Phase II Trial to Study the Tolerability and the Effectiveness of Imatinib in Patients With Chronic Myelogenous Leukemia in Chronic Phase in Relapse After Allogeneic Stem Cell Transplantation
Brief Title: Safety and Efficacy of Imatinib in Chronic Myelogenous Patients in Relapse After Stem Cell Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Collaborators: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 020947; CSTI571AFR05
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2005-09

CONDITIONS: Chronic Myeloid Leukemia
Keywords: CML; Imatinib mesylate; Stem cell transplantation
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: Imatinib mesylate

SUMMARY:
The aim of this phase II trial is asses the tolerability and the effectiveness of imatinib in patients with chronic myelogenous leukemia in chronic phase who are in relapse after stem cell transplantation.

DETAILED DESCRIPTION:
Patients will received Imatinib at a dose of 400mg daily. The tolerability of Imatinib given at a daily dose of 400mg will be assessed. The hematologic, cytogenetic and molecular responses will be evaluated at various check points.

Donor/recipient chimerism during Imatinib therapy will be assessed. Survival will be estimated.

ELIGIBILITY:
Inclusion Criteria:

* CML Ph+ (assessed by cytogenetic or FISH)
* Age ≥ 18 year at inclusion
* PS grade 0 to 2 (ECOG)
* previous allogeneic stem cell transplantation
* molecular, cytogenetic or haematological relapse in chronic phase after transplantation
* Immune therapy for graft versus host disease stopped within 2 months from inclusion
* Adequate and organ function, defined as the following: total bilirubin <3x uln, sgpt <3x uln, creatinine <2x uln.
* informed consent sign up

Exclusion Criteria:

* Age less than 18 y
* accelerated or blastic phase
* previous therapy with imatinib
* active malignancy other than CML or non-melanoma cancer of the skin
* current treatment with another investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2002-05; Study Completion 2007-07

PRIMARY OUTCOMES:
- to assess the tolerability of Imatinib given at a daily dose of 400mg
- to evaluate the hematologic, cytogenetic and molecular responses at various check points.

SECONDARY OUTCOMES:
- to assess donor/recipient chimerism during Imatinib therapy
- to evaluate the survival

CONTACTS AND LOCATIONS:
Overall Officials: François GUILHOT, MD, Study Chair — Department of Oncology Hematology and Cell therapy, University Hospital , 86021 Poitiers - FRANCE; Agnès DEVERGIE, MD, Principal Investigator — University Hospital "Saint-Louis" - Department of Hematology and Oncology - 75475 PARIS Cedex 10 (FRANCE)
Locations (1):
- University Hospital, Poitiers, France